CLINICAL TRIAL: NCT03121742
Title: A Pilot Study of a Smartphone-based Intervention for Suicidal Inpatients
Brief Title: A Study of a Smartphone-based Intervention for Suicidal Inpatients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Superseded by NCT03950765
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: American Psychological Foundation (Other); Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Evan M. Kleiman, Ph.D., Research Associate, Harvard University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB17-0483
Record Dates: First submitted 2017-04-06; First posted 2017-04-20 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Suicide, Attempted; Suicidal Ideation; Hopeless
Keywords: Suicide
MeSH Terms: conditions — Suicide, Attempted; Suicidal Ideation; Suicide | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as usual [TAU] plus assessment (Placebo Comparator): Patients will receive standard care plus assessment.
  Interventions: Behavioral: Treatment as Usual
- Treatment as usual [TAU] plus intervention (Experimental): Patients will receive standard care plus an ecological momentary intervention.
  Interventions: Behavioral: Ecological Momentary Intervention; Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Ecological Momentary Intervention — Patients will be taught four therapeutic intervention skills based on positive psychology and cognitive behavioral therapy. They will then be prompted to complete these interventions on a smartphone four times per day (and as needed) for the duration of their inpatient care and for 28 days afterwards.
  Arms: Treatment as usual [TAU] plus intervention
Behavioral: Treatment as Usual — Standard care as part of inpatient hospitalization.

SUMMARY:
Suicide is the most common form of deadly violence. Indeed, since more than 40,000 people die by suicide each year, people are 2.5 times more likely to die by their own hand than someone else's. The four weeks after discharge from inpatient care is an especially dangerous period in terms of suicide risk, possibly because of poor post-discharge treatment adherence and poor treatment efficacy during a suicide crisis. To reduce suicide risk both in general and during the post-discharge period, interventions are needed that (1) are easily adhered to and (2) are effective during a suicide crisis. The goal of the study is to pilot-test a suite of five smartphone-based ecological momentary interventions (EMI) that can be easily used during a suicide crisis. Two target hopelessness, two target loneliness, and one targets negative automatic thoughts associated with hopelessness and loneliness. Although these interventions are new to the study of suicide, they are all grounded in decades of empirical work and adapted from effective interventions in areas relating to suicide.

Participants will be 20 inpatients (n = 10 each in treatment as usual [TAU] plus intervention and TAU plus assessment [i.e., control] groups) from the Massachusetts General Hospital Inpatient Psychiatric Service. The investigators hypothesize that those in the TAU plus intervention group will have lower levels of suicidal ideation during the inpatient and post-discharge period than those in the TAU plus assessment group.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria include a recent (i.e., was included as the reason for admission) suicide attempt or serious suicidal ideation (i.e., ideation with at least 50% intent, assessed through either an explicit mention in the intake summary of intent greater than 50% or through this intent being inferred by clinical staff or in the notes [for example, if the patient notes they wanted to die more than they did not want to die during the attempt or episode of suicidal ideation]), English fluency, and access to an internet-capable smartphone (e.g., iPhone or Android).

Exclusion Criteria:

* Exclusion criteria include any factor that impairs the ability to effectively participate in the study (e.g., intellectual abilities that are too low to understand the study and/or consent process) or a diagnosis of any schizophrenia-spectrum or psychotic disorder.
* Additionally, patients who are on involuntary hospitalization status will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
Momentary Suicidal Ideation | Through study completion: ~35 days (7 days inpatient + 28 days post-discharge)
  Suicidal ideation as assessed by the ecological momentary assessment/intervention using a three item assessment of suicidal ideation that assess: (1) the desire to die by suicide, (2) the intention to die by suicide, and (3) the ability to resist the urge to die by suicide. This assessment will be given at four random times per day, as well as any time the participant initiates the survey or assessment.
Suicidal ideation | Through study completion: ~35 days (7 days inpatient + 28 days post-discharge)
  The occurrence of suicidal ideation (present/absent) over the course of the study, as assessed by the self-report version of the Self-Injurious Thoughts and Behaviors Interview (SITBI), administered at the end of the study.
Suicide attempts | Through study completion: ~35 days (7 days inpatient + 28 days post-discharge)
  The occurrence of suicide attempts (present/absent) over the course of the study, as assessed by the self-report version of the Self-Injurious Thoughts and Behaviors Interview (SITBI), administered at the end of the study.

SECONDARY OUTCOMES:
Hopelessness | Through study completion: ~35 days (7 days inpatient + 28 days post-discharge)
  Hopelessness as assessed by the ecological momentary assessment/intervention item with the heading "how are you feeling RIGHT NOW", with the label "hopeless" and options ranging from (1) not at all to (5) very much. This assessment will be given at four random times per day, as well as any time the participant initiates the survey or assessment.
Loneliness | Through study completion: ~35 days (7 days inpatient + 28 days post-discharge)
  Loneliness as assessed by the ecological momentary assessment/intervention item with the heading "how are you feeling RIGHT NOW", with the label "lonely" and options ranging from (1) not at all to (5) very much. This assessment will be given at four random times per day, as well as any time the participant initiates the survey or assessment.

IPD SHARING:
Plan to Share IPD: Undecided